CLINICAL TRIAL: NCT02874807
Title: Effects of the SGLT2-inhibitor Empagliflozin on Patients With SIADH - the SAND Study
Acronym: SAND
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAND study
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: SIADH
Keywords: Hyponatremia; SGLT2 inhibitor
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empagliflozin (Active Comparator): Treatment with empagliflozin 25mg once daily for four days
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Treatment with Placebo once daily for four days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin
  Arms: Empagliflozin
Other: Placebo
  Arms: Placebo

SUMMARY:
Syndrome of inappropriate antidiuresis (SIADH) is characterized by an imbalance of antidiuretic vasopressin (AVP) secretion. The impaired AVP regulation leads to water retention and secondary natriuresis and is a common cause for hyponatremia.

The therapeutic options, aside from treating the underlying disease, depend upon the onset and severity of the symptoms and involve usually fluid restriction or hypertonic saline infusion. Alternative therapeutic options are loop diuretics, administration of oral urea or vasopressin receptor antagonists (vaptans). Despite those options, there are a considerable number of patients which do not sufficiently respond, making additional therapy necessary.

Empagliflozin (Jardiance)® is a sodium glucose co-transporter 2 (SGLT2)-inhibitor, which is a new treatment option developed for patients with diabetes mellitus type 2. The SGLT2 is expressed in the proximal tubule and reabsorbs approximately 90 percent of the filtered glucose. The inhibition of SGLT2 results in renal excretion of glucose with subsequent osmotic diuresis. This mechanism could result in a therapeutic effect in patients with hypotonic hyponatremia as in SIADH.

The aim of this study is to evaluate whether empagliflozin (Jardiance)® has an effect on the serum sodium levels of patients with SIADH.

ELIGIBILITY:
Inclusion Criteria:

- Hyponatremia <130mmol/l due to SIADH

Exclusion Criteria:

* any Treatment for SIADH during >48h before study start
* severe illness with ICU-Admission
* Treatment with 3% sodium Chloride (NaCl) solution
* uncontrolled hypothyroidism
* uncontrolled adrenal insufficiency
* severe renal impairment (GFR <30ml/min), end stage renal disease
* severe hepatic impairment (Child-Pugh class C)
* systolic blood pressure <90mmHg
* Diabetes mellitus type 1
* acute myocardial infarction or chronic venous insufficiency (CVI)
* Treatment with SGLT2 Inhibitor, Lithium Chloride or Urea
* recurrent urinary-/genital tract infections
* contraindication for lowering blood pressure
* severe immunosuppression
* pregnancy or breastfeeding
* palliative care

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Serum sodium | 4 days
  The primary outcome is the change in serum sodium concentration from baseline to day 5, i.e. 4 days after start of treatment with study drug

SECONDARY OUTCOMES:
Serum sodium | 1 day
  Serum sodium concentration 1 day after start of Treatment with study drug
Serum sodium | 2 days
  Serum sodium concentration 2 days after start of treatment with study drug
Serum sodium | between day 1 to day 30
  Serum sodium concentration at discharge from hospital
Serum sodium | 30 days
  Serum sodium concentration 30 days after start of treatment with study drug
Fluid intake | 4 days
  amount of daily fluid intake
Urinary excretion | 4 days
  amount of daily urinary excretion
Serum electrolytes | 4 days
  change of serum electrolytes from baseline to day 5
Urinary electrolytes | 4 days
  Change of Serum electrolytes from baseline to day 5
Serum osmolality | 4 days
  Change of Serum osmolality from baseline to day 5
Urine osmolality | 4 days
  Change of urinary osmolality from baseline to day 5
Serum glucose | 4 days
  Change of Serum glucose from baseline to day 5
Urinary glucose | 4 days
  Change of urinary Glucose from baseline to day 5
Copeptin | 4 days
  Change of Copeptin from baseline to day 5
Aldosterone | 4 days
  Change of Aldosterone from baseline to day 5
Renin | 4 days
  Change of Renin from baseline to day 5
atrial natriuretic peptide (ANP) | 4 days
  Change of ANP from baseline to day 5
Brain-Natriuretic-Peptide (BNP) | 4 days
  Change of BNP from baseline to day 5
General well-being | 4 days
  course of General well-being from baseline to day 5 as assessed by patient's self-rating score
General well-being | 30 days
  course of General well-being from baseline to day 30 as assessed by patient's self-rating score
Symptoms of hyponatremia | 4 days
  course of hyponatremia symptoms from baseline to day 5
Symptoms of hyponatremia | 30 days
  Course of hyponatremia symptoms from baseline to day 30
Body weight | 4 days
  Change of Body weight from baseline to day 5
Blood pressure | 4 days
  Change of blood pressure from baseline to day 5
Heart rate | 4 days
  Change of heart rate from baseline to day 5
length of hospital stay | 30 days
  length of hospital stay
Treatment escalation | 30 days
  rate of Need for Treatment escalation
ICU Admission rate | 30 days
  rate of Admission to ICU
Recurrence hyponatremia | 30 days
  recurrence rate hyponatremia
Hospital readmission rate | 30 days
  rate of readmission

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof., MD, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nobbenhuis R, Refardt J, Vogt D, Sailer CO, Winzeler B, Christ-Crain M. Can treatment response to SGLT2-inhibitors in syndrome of inappropriate antidiuresis be predicted by copeptin, natriuretic peptides and inflammatory markers? Biomarkers. 2021 Nov;26(7):647-655. doi: 10.1080/1354750X.2021.1970808. Epub 2021 Aug 30. PMID 34412521